CLINICAL TRIAL: NCT07073690
Title: Real-World Treatment Patterns and Outcomes of Luspatercept in Patients With Lower-risk Myelodysplastic Syndromes (LR-MDS) in China ('REACH' Study)
Brief Title: Treatment Patterns and Outcomes in Patients With Lower-risk Myelodysplastic Syndromes Treated With Luspatercept in China
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA056-1166
Record Dates: First submitted 2025-07-10; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Myelodysplastic Syndromes
Keywords: Lower Risk Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — luspatercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants receiving luspatercept treatment
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — According to the product label

SUMMARY:
The purpose of this study is to evaluate the treatment patterns and clinical outcomes in adults with lower-risk MDS (LR-MDS) who were erythropoiesis-stimulating agents (ESA)-naïve and received luspatercept treatment in China

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 18 years of age.
* Documented diagnosis of no del(5q) MDS that meets lower-risk Myelodysplastic Syndromes (MDS) classification. (Diagnosis criteria and risk classification criteria are based on clinical practice)
* Patients who were erythropoiesis-stimulating agent (ESA)-naïve have received luspatercept monotherapy at least 2 cycles regardless of RS status.
* Historical documentation of anemia before luspatercept treatment.

Exclusion Criteria:

* Had a history of acute myeloid leukemia (AML) prior to MDS diagnosis.
* Received stem cell transplant prior to luspatercept treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise of individuals ≥18 years of age diagnosed with Lower-Risk Myelodysplastic Syndromes (LR-MDS) were erythropoiesis-stimulating agents (ESA)-naïve and received luspatercept treatment in China
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2025-11-26 (Estimated); Study Completion 2025-11-26 (Estimated)

PRIMARY OUTCOMES:
Participant red blood cell transfusion independence | Up to 12-weeks
Participants mean hemoglobin (Hb) increase ≥1.5 g/dL | Up to 12-weeks

SECONDARY OUTCOMES:
Participant transfusion independence and increase in hemoglobin (Hb) | Up to 48 weeks
Duration of luspatercept monotherapy treatment | Up to 48 weeks
Health Care Resource Utilization (HCRU) | Up to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Zhijian Xiao, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts